CLINICAL TRIAL: NCT02864914
Title: Post-authorisation Safety Study in Patients With Type 2 Diabetes Mellitus to Assess the Risk of Acute Liver Injury, Acute Kidney Injury and Chronic Kidney Disease, Severe Complications of Urinary Tract Infection, Genital Infections, and Diabetic Ketoacidosis Among Patients Treated With Empagliflozin Compared to Patients Treated With DPP-4 Inhibitors
Brief Title: Post-authorisation Safety Study in Patients With Type 2 Diabetes to Assess the Risk of Liver Injury, Kidney Injury, Urinary Tract and Genital Infections, and Diabetic Ketoacidosis in Patients Treated With Empagliflozin, Compared to DPP-4 Inhibitors
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245.96
Record Dates: First submitted 2016-05-13; First posted 2016-08-12 (Estimated); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Empagliflozin: All eligible patients type 2 diabetes mellitus initiating Empagliflozin treatment within the study period, from existing data of routine medical care in the Clinical Practice Research Datalink (CPRD) in the United Kingdom (UK), HealthCore Integrated Research Database (HIRD) in the United States (US), and Danish Population Registries (Danish Registries) in Denmark.
  The study period started on 01 August 2014, the date of empagliflozin launch in the UK, US, and Denmark. The study end date was 01 August 2019 in CPRD and Danish Registries and 31 July 2019 in HIRD.
  Interventions: Drug: Empagliflozin
- DPP-4 inhibitors: All eligible patients with type 2 diabetes mellitus initiating Dipeptidyl peptidase-4 (DPP-4) inhibitors treatment within the study period, existing data of routine medical care in the Clinical Practice Research Datalink (CPRD) in the United Kingdom (UK), HealthCore Integrated Research Database (HIRD) in the United States (US), and Danish Population Registries (Danish Registries) in Denmark.
  The study period started on 01 August 2014, the date of empagliflozin launch in the UK, US, and Denmark. The study end date was 01 August 2019 in CPRD and Danish Registries and 31 July 2019 in HIRD.
  Interventions: Drug: DPP-4 inhibitors

INTERVENTIONS:
Drug: Empagliflozin — drug
  Groups: Empagliflozin
Drug: DPP-4 inhibitors — drug
  Groups: DPP-4 inhibitors

SUMMARY:
Empagliflozin (Jardiance), a highly potent and selective inhibitor of the sodium-glucose cotransporter 2 (SGLT2), was approved in Europe in May 2014 for the treatment of type 2 diabetes mellitus (T2DM) to improve glycaemic control in adults. As part of the risk management plan, Boehringer Ingelheim International GmbH (BI) has committed to conduct a post-authorisation safety study (PASS) to evaluate the liver and renal safety of empagliflozin. The study will also evaluate the risks of severe complications of urinary tract infections (UTIs) and genital infections. To evaluate the association between empagliflozin use and mentioned outcomes routinely collected health information from the Clinical Practice Research Datalink (CPRD), the Hospital Episodes Statistics, and Office of National Statistic will be used. This PASS will be conducted through an observational cohort study among adult patients with T2DM and at least 12 months of continuous enrolment in the CPRD where new users of empagliflozin will be compared to new users of dipeptidyl peptidase-4 (DPP4) inhibitors. Estimations will be made on the crude and adjusted incidence rates and adjusted incidence rate ratios of the primary and secondary outcomes.

ELIGIBILITY:
Inclusion criteria:

* Patients will have T2DM, be initiating treatment with a study medication, and have at least 12 months of continuous registration in CPRD.
* Further inclusion criteria apply

Exclusion criteria:

* Patients will not have T1DM, will have no prior use of an SGLT2 inhibitor or DPP4 inhibitor, and will not be initiating a SGLT2-DPP4 fixed-dose combination.
* Additional different exclusion criteria will be applied according to each outcomes of interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2DM eligible patients in CPRD
Sampling Method: Non-Probability Sample
Enrollment: 333580 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- RTI health solutions, One Or Multiple Sites, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional observational cohort study using existing data from routine medical care in the Clinical Practice Research Datalink in the United Kingdom, the Danish Population Registries in Denmark, and the HealthCore Integrated Research Database in the United States investigating safety among patients with type 2 diabetes mellitus treated with empagliflozin versus Dipeptidyl peptidase-4 inhibitors.
Pre-assignment Details: All subjects were screened for eligibility to ensure that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
Period: Overall Study
Arm/Group | Empagliflozin | DPP-4 Inhibitors
Started | 76174 | 257406
Propensity Score-trimmed Cohort for DKA (The propensity score (PS)-trimmed cohort was created by trimming extreme values of PS from a Diabetic ketoacidosis (DKA)-specific PS model including all DKA-related variables.) | 64599 | 203315
Propensity Score-trimmed Cohort for AKI (The propensity score (PS)-trimmed cohort was created by trimming extreme values of PS from a acute kidney injury (AKI)-specific PS model including all AKI-related variables.) | 58393 | 167823
Propensity Score-trimmed Cohort for ALI2 (The propensity score (PS)-trimmed cohort was created by trimming extreme values of PS from a Acute liver injury with or without predisposing conditions (ALI2)-specific PS model including all ALI2-related variables.) | 62917 | 197172
Propensity Score-trimmed Cohort for CKD - CPRD Only (The propensity score (PS)-trimmed cohort was created by trimming extreme values of PS from a Chronic kidney disease (CKD)-specific PS model including all CKD-related variables. CKD was evaluated only in CPRD database.) | 13256 | 62435
Propensity Score-trimmed Cohort for GIM - CPRD Only (The propensity score (PS)-trimmed cohort in males was created by trimming extreme values of PS from a genital infection in males (GIM)-specific PS model including all GIM-related variables. GIM was evaluated only in CPRD database.) | 8272 | 45683
Propensity Score-trimmed Cohort for UTI - CPRD Only (The propensity score (PS)-trimmed cohort was created by trimming extreme values of PS from a Urinary tract infection (UTI)-specific PS model including all UTI-related variables. UTI was evaluated only in CPRD database.) | 14050 | 77330
Propensity Score-trimmed Cohort for GIF - CPRD Only (The propensity score (PS)-trimmed cohort in females was created by trimming extreme values of PS from a genital infection in females (GIF)-specific PS model including all GIF-related variables. GIF was evaluated only in CPRD database.) | 5802 | 31904
Propensity Score-trimmed Cohort for ALI1 (The propensity score (PS)-trimmed cohort was created by trimming extreme values of PS from a Acute liver injury with no predisposing conditions (ALI1)-specific PS model including all ALI1-related variables. The number of participants from the Danish Registries treated with empagliflozin, and treated with DPP-4 inhibitors and ≥ 3 glucose-lowering drugs are not reported due to the Danish small cell count policy.) | 36053 | 154554
Completed | 76174 | 257406
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible subjects who strictly met all inclusion and none of the exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin | DPP-4 Inhibitors | Total
Number analyzed (Participants) | 76174 | 257406 | 333580
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (10.8) | 62.1 (13.1) | 61.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30774 | 110654 | 141428
  Male | 45400 | 146752 | 192152
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rates of Acute Liver Injury (ALI) in Patients With no Predisposing Conditions (ALI1) in Propensity Score-trimmed Cohort for ALI1
Description: Incidence rates (IRs) of acute liver injury (ALI) in patients with no predisposing conditions (ALI1) in propensity score-trimmed study cohorts for ALI1 are reported.
  Unadjusted IRs were computed as the number of events divided by the total person-years at risk in the empagliflozin and DPP-4 inhibitors cohorts overall and for subgroups with and without insulin use at the index date. IRs adjusted for propensity score decile were generated for empagliflozin and DPP-4 inhibitor cohorts overall (not stratified by any other variable). These estimates with corresponding 95% confidence interval (CIs) were generated using a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model.
Time Frame: up to 5 years
Population: All eligible subjects who strictly met all inclusion and none of the exclusion criteria, and with non-missing ALI results and with no predisposing conditions (ALI1) were included. The cohort after propensity score trimming (extreme values of propensity score were trimmed) was used. A ALI1-specific propensity score model was used for the propensity score including all ALI1-related variables. Due to the Danish small cell count policy, some cohorts were not reported (see limits & caveats).
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Groups:
- Empagliflozin - CPRD (After Propensity Score Trimming): All eligible patients with type 2 diabetes mellitus initiating Empagliflozin treatment within the study period, existing data of routine medical care in the Clinical Practice Research Datalink (CPRD) in the United Kingdom (UK).
  This group includes all eligible participants initiating Empagliflozin after propensity score-trimming, where the model used for propensity score was endpoint-specific including all variables related to the endpoint.
- Empagliflozin - HIRD (After Propensity Score Trimming): All eligible patients with type 2 diabetes mellitus initiating Empagliflozin treatment within the study period, existing data of routine medical care in the HealthCore Integrated Research Database (HIRD) in the United States (US).
  This group includes all eligible participants initiating Empagliflozin after propensity score-trimming, where the model used for propensity score was endpoint-specific including all variables related to the endpoint.
- DPP-4 Inhibitors - CPRD (After Propensity Score Trimming): All eligible patients with type 2 diabetes mellitus initiating Dipeptidyl peptidase-4 (DPP-4) inhibitors treatment within the study period, existing data of routine medical care in the Clinical Practice Research Datalink (CPRD) in the United Kingdom (UK).
  This group includes all eligible participants initiating DPP-4 inhibitors after propensity score-trimming, where the model used for propensity score was endpoint-specific including all variables related to the endpoint.
- DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming): All eligible patients with type 2 diabetes mellitus initiating Dipeptidyl peptidase-4 (DPP-4) inhibitors treatment within the study period with <3 glucose-lowering drugs, existing data of routine medical care in the Danish Population Registries (Danish Registries) in Denmark.
  This group includes all eligible participants initiating DPP-4 inhibitors after propensity score-trimming, where the model used for propensity score was endpoint-specific including all variables related to the endpoint.
- DPP-4 Inhibitors - HIRD (After Propensity Score Trimming): All eligible patients with type 2 diabetes mellitus initiating Dipeptidyl peptidase-4 (DPP-4) inhibitors treatment within the study period, existing data of routine medical care in the HealthCore Integrated Research Database (HIRD) in the United States (US).
  This group includes all eligible participants initiating DPP-4 inhibitors after propensity score-trimming, where the model used for propensity score was endpoint-specific including all variables related to the endpoint.
Arm/Group | Empagliflozin - CPRD (After Propensity Score Trimming) | Empagliflozin - HIRD (After Propensity Score Trimming) | DPP-4 Inhibitors - CPRD (After Propensity Score Trimming) | DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) | DPP-4 Inhibitors - HIRD (After Propensity Score Trimming)
Number analyzed (Participants) | 11189 | 24864 | 61254 | 27404 | 65896
Events per 1000 person-years | 0.60 [0.27 to 1.36] | 1.21 [0.79 to 1.86] | 1.09 [0.75 to 1.59] | NA [NA to NA] — Due to the low number of events, the Poisson regression models had convergence/validity issues. Therefore, results were reported as "not estimable". | 1.41 [1.04 to 1.92]
Statistical Analysis 1: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs Empagliflozin - HIRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - HIRD (After Propensity Score Trimming); Adjusted IR ratio was generated overall with corresponding 95% CIs through the application of a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model; Test type: Other; Adjusted incidence rate ratio = 0.77, 95% CI 2-sided [0.50 to 1.19] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 2: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.55, 95% CI 2-sided [0.23 to 1.32] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 3: Comparison: Empagliflozin - HIRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - HIRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.86, 95% CI 2-sided [0.52 to 1.41] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors

2. Primary Outcome: Incidence Rates of Acute Kidney Injury (AKI) in Propensity Score-trimmed Cohort for AKI
Description: Incidence rates (IRs) of acute kidney injury (AKI) in propensity score-trimmed cohort for AKI are reported.
  Unadjusted IRs were computed as the number of events divided by the total person-years at risk in the empagliflozin and DPP-4 inhibitors cohorts overall and for subgroups with and without insulin use at the index date. IRs adjusted for propensity score decile were generated for empagliflozin and DPP-4 inhibitor cohorts overall (not stratified by any other variable). These estimates with corresponding 95% CIs were generated through the application of a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model.
Time Frame: up to 5 years
Population: All eligible subjects who strictly met all inclusion and none of the exclusion criteria. The cohort after propensity score trimming (extreme values of propensity score were trimmed) was used. A AKI-specific propensity score model was used for the propensity score including all AKI-related variables.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Groups:
- Empagliflozin - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming): All eligible patients with type 2 diabetes mellitus initiating Empagliflozin treatment within the study period with <3 glucose-lowering drugs, existing data of routine medical care in the Danish Population Registries (Danish Registries) in Denmark.
  This group includes all eligible participants initiating Empagliflozin after propensity score-trimming, where the model used for propensity score was endpoint-specific including all variables related to the endpoint.
- Empagliflozin - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming): All eligible patients with type 2 diabetes mellitus initiating Empagliflozin treatment within the study period with ≥3 glucose-lowering drugs, existing data of routine medical care in the Danish Population Registries (Danish Registries) in Denmark.
  This group includes all eligible participants initiating Empagliflozin after propensity score-trimming, where the model used for propensity score was endpoint-specific including all variables related to the endpoint.
- DPP-4 Inhibitors - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming): All eligible patients with type 2 diabetes mellitus initiating Dipeptidyl peptidase-4 (DPP-4) inhibitors treatment within the study period with ≥3 glucose-lowering drugs, existing data of routine medical care in the Danish Population Registries (Danish Registries) in Denmark.
  This group includes all eligible participants initiating DPP-4 inhibitors after propensity score-trimming, where the model used for propensity score was endpoint-specific including all variables related to the endpoint.
Arm/Group | Empagliflozin - CPRD (After Propensity Score Trimming) | Empagliflozin - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) | Empagliflozin - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming) | Empagliflozin - HIRD (After Propensity Score Trimming) | DPP-4 Inhibitors - CPRD (After Propensity Score Trimming) | DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) | DPP-4 Inhibitors - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming) | DPP-4 Inhibitors - HIRD (After Propensity Score Trimming)
Number analyzed (Participants) | 13215 | 9296 | 5362 | 30520 | 61879 | 28897 | 2297 | 74750
Events per 1000 person-years | 4.64 [3.51 to 6.12] | 3.41 [2.31 to 5.02] | 2.60 [1.54 to 4.40] | 10.96 [9.61 to 12.49] | 11.43 [10.21 to 12.79] | 4.96 [4.17 to 5.89] | 6.31 [3.40 to 11.71] | 16.89 [15.56 to 18.33]
Statistical Analysis 1: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs Empagliflozin - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) vs Empagliflozin - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming) vs Empagliflozin - HIRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) vs DPP-4 Inhibitors - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming) vs DPP-4 Inhibitors - HIRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.54, 95% CI 2-sided [0.41 to 0.73] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 2: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.41, 95% CI 2-sided [0.30 to 0.55] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 3: Comparison: Empagliflozin - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) vs DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.69, 95% CI 2-sided [0.45 to 1.05] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 4: Comparison: Empagliflozin - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming) vs DPP-4 Inhibitors - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.41, 95% CI 2-sided [0.20 to 0.86] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 5: Comparison: Empagliflozin - HIRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - HIRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.65, 95% CI 2-sided [0.56 to 0.76] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors

3. Primary Outcome: Incidence Rates of Diabetic Ketoacidosis (DKA) in Propensity Score-trimmed Cohort for DKA
Description: Incidence rates (IRs) of diabetic ketoacidosis (DKA) in propensity score-trimmed cohort for DKA are reported.
  Unadjusted IRs were computed as the number of events divided by the total person-years at risk in the empagliflozin and DPP-4 inhibitors cohorts overall and for subgroups with and without insulin use at the index date. IRs adjusted for propensity score decile were generated for empagliflozin and DPP-4 inhibitor cohorts overall (not stratified by any other variable). These estimates with corresponding 95% CIs were generated through the application of a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model.
Time Frame: up to 5 years
Population: All eligible subjects who strictly met all inclusion and none of the exclusion criteria. The cohort after propensity score trimming (extreme values of propensity score were trimmed) was used. A DKA-specific propensity score model was used for the propensity score including all DKA-related variables.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Empagliflozin - CPRD (After Propensity Score Trimming) | Empagliflozin - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) | Empagliflozin - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming) | Empagliflozin - HIRD (After Propensity Score Trimming) | DPP-4 Inhibitors - CPRD (After Propensity Score Trimming) | DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) | DPP-4 Inhibitors - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming) | DPP-4 Inhibitors - HIRD (After Propensity Score Trimming)
Number analyzed (Participants) | 14086 | 9923 | 5905 | 34685 | 77408 | 33973 | 2742 | 89192
Events per 1000 person-years | 2.57 [1.78 to 3.70] | 1.50 [0.85 to 2.64] | NA [NA to NA] — Due to the low number of events, the Poisson regression models had convergence/validity issues. Therefore, results were reported as "not estimable". | 3.62 [2.93 to 4.48] | 0.92 [0.67 to 1.28] | 0.70 [0.46 to 1.07] | NA [NA to NA] — Due to the low number of events, the Poisson regression models had convergence/validity issues. Therefore, results were reported as "not estimable". | 1.82 [1.47 to 2.26]
Statistical Analysis 1: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs Empagliflozin - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) vs Empagliflozin - HIRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) vs DPP-4 Inhibitors - HIRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 2.19, 95% CI 2-sided [1.74 to 2.76] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 2: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 2.78, 95% CI 2-sided [1.77 to 4.36] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 3: Comparison: Empagliflozin - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) vs DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 2.14, 95% CI 2-sided [1.11 to 4.12] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 4: Comparison: Empagliflozin - HIRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - HIRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 1.99, 95% CI 2-sided [1.48 to 2.66] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors

4. Primary Outcome: Incidence Rates of Severe Complications of Urinary Tract Infections (UTIs) in Propensity Score-trimmed Cohort for UTI - CPRD Only
Description: Incidence rates (IRs) of severe complications of urinary tract infections (UTIs) in propensity score-trimmed cohort for UTI among CPRD participants are reported.
  Unadjusted IRs were computed as the number of events divided by the total person-years at risk in the empagliflozin and DPP-4 inhibitors cohorts overall and for subgroups with and without insulin use at the index date. IRs adjusted for propensity score decile were generated for empagliflozin and DPP-4 inhibitor cohorts overall (not stratified by any other variable). These estimates with corresponding 95% CIs were generated through the application of a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model.
Time Frame: up to 5 years
Population: All eligible subjects who strictly met all inclusion and none of the exclusion criteria. The cohort after propensity score trimming (extreme values of propensity score were trimmed) was used. A UTI-specific propensity score model was used for the propensity score including all UTI-related variables. Because UTI was evaluated only in CPRD database, only participants from CPRD were used.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Empagliflozin - CPRD (After Propensity Score Trimming) | DPP-4 Inhibitors - CPRD (After Propensity Score Trimming)
Number analyzed (Participants) | 14050 | 77330
Events per 1000 person-years | 3.32 [2.42 to 4.54] | 6.47 [5.64 to 7.42]
Statistical Analysis 1: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.51, 95% CI 2-sided [0.37 to 0.72] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors

5. Primary Outcome: Incidence Rates of Genital Infections in Males (GIM) in Propensity Score-trimmed Cohort for GIM - CPRD Only
Description: Incidence rates (IRs) of genital infections in males (GIM) in propensity score-trimmed cohorts for GIM among CPRD participants are reported.
  Unadjusted IRs were computed as the number of events divided by the total person-years at risk in the empagliflozin and DPP-4 inhibitors cohorts overall and for subgroups with and without insulin use at the index date. IRs adjusted for propensity score decile were generated for empagliflozin and DPP-4 inhibitor cohorts overall (not stratified by any other variable). These estimates with corresponding 95% CIs were generated through the application of a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model.
Time Frame: up to 5 years
Population: All eligible subjects who strictly met all inclusion and none of the exclusion criteria. The cohort after propensity score trimming (extreme values of propensity score were trimmed) was used. A GIM-specific propensity score model was used for the propensity score including all GIM-related variables. Because genital infection was evaluated only in CPRD database, only participants from CPRD were used.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Empagliflozin - CPRD (After Propensity Score Trimming) | DPP-4 Inhibitors - CPRD (After Propensity Score Trimming)
Number analyzed (Participants) | 8272 | 45683
Events per 1000 person-years | 47.23 [42.28 to 52.76] | 11.70 [10.45 to 13.10]
Statistical Analysis 1: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 4.04, 95% CI 2-sided [3.46 to 4.71] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors

6. Primary Outcome: Incidence Rates of Genital Infections in Females (GIF) in Propensity Score-trimmed Cohort for GIF - CPRD Only
Description: Incidence rates (IRs) of genital infections in females (GIF) in propensity score-trimmed cohort for GIF among CPRD participants are reported.
  Unadjusted IRs were computed as the number of events divided by the total person-years at risk in the empagliflozin and DPP-4 inhibitors cohorts overall and for subgroups with and without insulin use at the index date. IRs adjusted for propensity score decile were generated for empagliflozin and DPP-4 inhibitor cohorts overall (not stratified by any other variable). These estimates with corresponding 95% CIs were generated through the application of a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model.
Time Frame: up to 5 years
Population: All eligible subjects who strictly met all inclusion and none of the exclusion criteria. The cohort after propensity score trimming (extreme values of propensity score were trimmed) was used. A GIF-specific propensity score model was used for the propensity score including all GIF-related variables. Because genital infection was evaluated only in CPRD database, only participants from CPRD were used.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Empagliflozin - CPRD (After Propensity Score Trimming) | DPP-4 Inhibitors - CPRD (After Propensity Score Trimming)
Number analyzed (Participants) | 5802 | 31940
Events per 1000 person-years | 79.65 [71.72 to 88.45] | 24.58 [22.28 to 27.13]
Statistical Analysis 1: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 3.24, 95% CI 2-sided [2.81 to 3.74] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors

7. Secondary Outcome: Incidence Rates of Acute Liver Injury (ALI) in Patients With or Without Predisposing Conditions (ALI2) in Propensity Score-trimmed Cohort for ALI2
Description: Incidence rates (IRs) of acute liver injury (ALI) in patients with or without predisposing conditions (ALI2) in propensity score-trimmed cohort for ALI2 are reported.
  Unadjusted IRs were computed as the number of events divided by the total person-years at risk in the empagliflozin and DPP-4 inhibitors cohorts overall and for subgroups with and without insulin use at the index date. IRs adjusted for propensity score decile were generated for empagliflozin and DPP-4 inhibitor cohorts overall (not stratified by any other variable). These estimates with corresponding 95% CIs were generated through the application of a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model.
Time Frame: up to 5 years
Population: All eligible subjects who strictly met all inclusion and none of the exclusion criteria. The cohort after propensity score trimming (extreme values of propensity score were trimmed) was used. A ALI2-specific propensity score model was used for the propensity score including all ALI2-related variables.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Empagliflozin - CPRD (After Propensity Score Trimming) | Empagliflozin - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) | Empagliflozin - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming) | Empagliflozin - HIRD (After Propensity Score Trimming) | DPP-4 Inhibitors - CPRD (After Propensity Score Trimming) | DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) | DPP-4 Inhibitors - Danish Registries ≥3 Glucose-lowering Drugs (After Propensity Score Trimming) | DPP-4 Inhibitors - HIRD (After Propensity Score Trimming)
Number analyzed (Participants) | 13913 | 9681 | 5740 | 33583 | 75580 | 33308 | 2661 | 85623
Events per 1000 person-years | 1.33 [0.81 to 2.19] | 1.23 [0.66 to 2.31] | NA [NA to NA] — Due to the low number of events, the Poisson regression models had convergence/validity issues. Therefore, results were reported as "not estimable". | 4.19 [3.43 to 5.11] | 2.67 [2.14 to 3.33] | 1.86 [1.43 to 2.41] | NA [NA to NA] — Due to the low number of events, the Poisson regression models had convergence/validity issues. Therefore, results were reported as "not estimable". | 5.47 [4.79 to 6.26]
Statistical Analysis 1: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs Empagliflozin - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) vs Empagliflozin - HIRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) vs DPP-4 Inhibitors - HIRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.70, 95% CI 2-sided [0.56 to 0.88] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 2: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.50, 95% CI 2-sided [0.29 to 0.85] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 3: Comparison: Empagliflozin - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming) vs DPP-4 Inhibitors - Danish Registries <3 Glucose-lowering Drugs (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.66, 95% CI 2-sided [0.34 to 1.29] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors
Statistical Analysis 4: Comparison: Empagliflozin - HIRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - HIRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.77, 95% CI 2-sided [0.61 to 0.97] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors

8. Secondary Outcome: Incidence Rates of Chronic Kidney Disease (CKD) in Propensity Score-trimmed Cohort for CKD - CPRD Only
Description: Incidence rates (IRs) of chronic kidney disease (CKD) in propensity score-trimmed cohort for CKD among CPRD participants are reported.
  Unadjusted IRs were computed as the number of events divided by the total person-years at risk in the empagliflozin and DPP-4 inhibitors cohorts overall and for subgroups with and without insulin use at the index date. IRs adjusted for propensity score decile were generated for empagliflozin and DPP-4 inhibitor cohorts overall (not stratified by any other variable). These estimates with corresponding 95% CIs were generated through the application of a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model.
Time Frame: up to 5 years
Population: All eligible subjects who strictly met all inclusion and none of the exclusion criteria. The cohort after propensity score trimming (extreme values of propensity score were trimmed) was used. A CKD-specific propensity score model was used for the propensity score including all CKD-related variables. Because CKD was evaluated only in CPRD database, only participants from CPRD were used.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Empagliflozin - CPRD (After Propensity Score Trimming) | DPP-4 Inhibitors - CPRD (After Propensity Score Trimming)
Number analyzed (Participants) | 13256 | 62435
Events per 1000 person-years | 9.32 [7.68 to 11.31] | 17.73 [16.16 to 19.45]
Statistical Analysis 1: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 0.53, 95% CI 2-sided [0.43 to 0.65] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors

9. Secondary Outcome: Incidence Rates of Severe Genital Infections in Males (GIMH) in Propensity Score-trimmed Cohort for GIM - CPRD Only
Description: Incidence rates (IRs) of severe genital infections in males (GIMH) in propensity score-trimmed cohort for GIM among CPRD participants are reported.
  Unadjusted IRs were computed as the number of events divided by the total person-years at risk in the empagliflozin and DPP-4 inhibitors cohorts overall and for subgroups with and without insulin use at the index date. IRs adjusted for propensity score decile were generated for empagliflozin and DPP-4 inhibitor cohorts overall (not stratified by any other variable). These estimates with corresponding 95% CIs were generated through the application of a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model.
Time Frame: up to 5 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Empagliflozin - CPRD (After Propensity Score Trimming) | DPP-4 Inhibitors - CPRD (After Propensity Score Trimming)
Number analyzed (Participants) | 8272 | 45683
Events per 1000 person-years | 43.35 [38.63 to 48.65] | 10.72 [9.53 to 12.07]
Statistical Analysis 1: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 4.04, 95% CI 2-sided [3.44 to 4.75] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors

10. Secondary Outcome: Incidence Rates of Severe Genital Infections in Females (GIFH) in Propensity Score-trimmed Cohort for GIF - CPRD Only
Description: Incidence rates (IRs) of severe genital infections in females (GIFH) in propensity score-trimmed cohort for GIF among CPRD participants are reported.
  Unadjusted IRs were computed as the number of events divided by the total person-years at risk in the empagliflozin and DPP-4 inhibitors cohorts overall and for subgroups with and without insulin use at the index date. IRs adjusted for propensity score decile were generated for empagliflozin and DPP-4 inhibitor cohorts overall (not stratified by any other variable). These estimates with corresponding 95% CIs were generated through the application of a Poisson regression model where the outcome was modelled as a function of treatment cohort (empagliflozin or DPP-4 inhibitors) and propensity score decile (specified as a categorical variable) with the log of time of exposure (in years) as the offset. If any variable remained unbalanced after trimming, it was added as an independent variable in the Poisson regression model.
Time Frame: up to 5 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years
Arm/Group | Empagliflozin - CPRD (After Propensity Score Trimming) | DPP-4 Inhibitors - CPRD (After Propensity Score Trimming)
Number analyzed (Participants) | 5802 | 31940
Events per 1000 person-years | 58.42 [51.73 to 65.97] | 17.48 [15.57 to 19.64]
Statistical Analysis 1: Comparison: Empagliflozin - CPRD (After Propensity Score Trimming) vs DPP-4 Inhibitors - CPRD (After Propensity Score Trimming); [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted incidence rate ratio = 3.34, 95% CI 2-sided [2.83 to 3.95] — Adjusted incidence rate ratio = incidence rate empagliflozin / incidence rate DPP-4 inhibitors

ADVERSE EVENTS:
Time Frame: No applicable.
Description: This study used existing data and adverse events were not planned to be collected and reported. The "0" in the All-cause Mortality, Serious Adverse Events, and Other Adverse Events sections below indicating "Not applicable".
Arm/Group | Empagliflozin | DPP-4 Inhibitors
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
In the outcome measure ALI1, the number of patients after trimming belonging to the Danish Registries and treated with Empagliflozin, as well as with DPP-4 inhibitors and ≥ 3 glucose-lowering drugs, cannot be reported since the number of events in Danish Registries was 1 to 4, and the total cannot be given to avoid back-calculation of values due to the Danish small cell count policy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT02864914/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT02864914/SAP_001.pdf